CLINICAL TRIAL: NCT00819325
Title: Prevention of Neointimal Proliferation With Aggressive Reduction of Glucose Concentrations (Pioglitazone) Study -- PPAR-G -- An IVUS Pilot Feasibility Study in Type 2 Diabetic Patients.
Brief Title: Prevention of Instent Renarrowing With Aggressive Glucose Lowering With Pioglitazone in Diabetic Patients
Acronym: PPAR-G
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen Elizabeth II Health Sciences Centre (Other)
Collaborators: Nova Scotia Health Research Foundation (Other Government)
Responsible Party: Lawrence Title, QE II Health Sciences Centre, Division of Cardiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NSHRF #404N-01; NSHRF grant #404N-01
Record Dates: First submitted 2009-01-06; First posted 2009-01-08 (Estimated); Last update posted 2009-01-08 (Estimated); Status verified 2009-01

CONDITIONS: Coronary Artery Disease; Angina Pectoris; Type 2 Diabetes Mellitus; Percutaneous Coronary Intervention
Keywords: diabetes; stents; restenosis; thiazolidinediones; coronary atherosclerosis
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Pioglitazone; Hypoglycemic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive glycemic control (Experimental): Included routine use of pioglitazone (30 mg/d) for 6 months in addition to titration of their other oral hypoglycemic agents in order to get the HbA1c<6%.
  Interventions: Drug: pioglitazone; Drug: oral hypoglycemic agents
- conservative glycemic control (Active Comparator): Included titration of oral hypoglycemic agents to get HbA1c<7% without the use of a thiazolidinedione.
  Interventions: Drug: oral hypoglycemic agents

INTERVENTIONS:
Drug: pioglitazone — pioglitazone 30mg p.o. once a day for 6 months
  Arms: Intensive glycemic control
Drug: oral hypoglycemic agents — sulfonylurea or metformin

SUMMARY:
Patients with diabetes have worse outcomes after percutaneous coronary intervention (PCI) procedures, compared to those patients without diabetes. They are at increased risk of death, heart attack, or needing further procedures due to renarrowing of their coronary narrowings after implantation of a coronary stent. Studies have suggested that poor control of diabetes may be partly responsible for these poor outcomes. Thiazolidinedione drugs, such as pioglitazone, can improve the diabetes control and make the patient more sensitive to the effects of insulin. Preliminary studies suggest that pioglitazone may also help prevent renarrowing after PCI.

This study was a pilot study designed to determine whether more aggressive treatment of the diabetes with the routine use of the drug pioglitazone (30mg/day for 6 months), in addition to the patient's usual diabetic medications adjusted to optimize their diabetic control (get glycated hemoglobin < 7%), could reduce the amount of tissue buildup within the stent after 6 months, compared to a group less aggressively treated without pioglitazone and their usual medications for diabetes.

An intravascular ultrasound probe was used to assess the extent of tissue buildup within the stent and this was performed immediately after the PCI as a baseline and repeated after 6 months of therapy.

The investigators hypothesize that the more aggressive diabetic treatment with pioglitazone would reduce the extent of tissue growth within the stent after 6 months of therapy.

DETAILED DESCRIPTION:
Background: Despite drug-eluting stents (DES), diabetic patients remain at high risk of restenosis and poor clinical outcomes after percutaneous coronary intervention (PCI). Studies have suggested poor glycemic control and insulin resistance may be predictors of poor outcomes after PCI. There are conflicting studies as to whether strategies to improve glycemic control can improve outcomes after PCI. Thiazolidinediones, such as pioglitazone (PIO), may have anti-restenotic benefits, independent of glycemic control.

Study design: This study was a single centre prospective, randomized, open-label, blinded-endpoint (PROBE) parallel design trial. Type 2 diabetic patients, treated with diet or oral antidiabetic medication (sulfonylurea vs. metformin or combination; but no thiazolidinedione or insulin), who are undergoing elective or urgent PCI with stenting were eligible. Fifty type 2 diabetic patients were randomly assigned to either: intensive glycemic control: pioglitazone (PIO; 30 mg/d x 6 months) in addition to titration of oral hypoglycemic agents (OHA) to get HbA1c<6% (PIO: n=25) vs. conservative glycemic control: titration of OHA to get HbA1c<7% (CONTROL: n=25). Intravascular ultrasound (IVUS) was performed immediately after PCI and repeated at 6 months to determine the effect on instent neointimal plaque volume and area. Coronary stenting was carried out in a standard fashion, with routine use of a glycoprotein 2b/3a inhibitor during the procedure. From August 2002 until June 2005, DES were not permitted in the protocol. After June 2005, we amended the protocol to allow DES, as they had become routinely used in diabetic patients in our institution, especially for vessel size <3mm and/or lesion length>15mm. DES were used in 7 PIO and 11 CONTROL subjects, and bare metal stents (BMS) in the rest. Patients were then followed with clinic visits at 1, 3 and 6 months. OHA, other than pioglitazone, were adjusted in a stepwise manner in order to attain the HbA1c targets. Other concomitant medications, including anti-anginals, lipid-lowering therapy, and antihypertensive medication were adjusted according to their clinical need and current Canadian guidelines. After 6 months treatment, or before if clinically indicated, all subjects were to return for repeat cardiac catheterization, including repeat coronary angiography and IVUS of the intervened vessel to assess the serial change in luminal dimensions. Fasting blood was collected for plasma glucose, HbA1c, insulin, lipid profile, hs-CRP, adiponectin, leptin, matrix metalloproteinase-9, and interleukin-6 at the time of PCI and at the follow-up IVUS. If the patient developed recurrent ischemic symptoms before 6 months, the final IVUS could be performed earlier, if they were found to have clinically-significant restenosis (diameter stenosis > 50%). Otherwise, patients were still encouraged to have their protocol 6 month IVUS follow-up. 41 patients (n=20 PIO, n=21 CONTROL) had analyzable pairs of IVUS.

Study hypothesis: We hypothesized that there would be significantly less instent neointimal proliferation on IVUS at 6 months in the group receiving aggressive glycemic control plus the thiazolidinedione pioglitazone. We also hypothesized that the reduction in neointimal hyperplasia will likely relate to improvements in glycemic control (HbA1c) and insulin resistance. Additionally, we wanted to explore the biochemical predictors (glucose parameters, lipids, inflammatory markers, adipokines) for neointimal proliferation.

ELIGIBILITY:
Inclusion Criteria:

* between the ages 30 to 80 years
* had type 2 diabetes mellitus treated with diet or oral hypoglycemic agents (OHA: sulfonylurea or metformin alone or the combination of sulfonylurea or metformin as long as metformin dose was < 2000 mg/d)
* All patients were undergoing either elective or urgent PCI of a de novo native coronary lesion (> 70 % diameter stenosis) in a vessel ≥ 2.5 mm diameter that was felt to be suitable for stenting and an IVUS examination.

Exclusion Criteria:

* left main > 50 % stenosis
* ongoing congestive heart failure or left ventricular ejection fraction < 30%
* primary PCI for ST elevation MI
* use of insulin or thiazolidinedione therapy (rosiglitazone or pioglitazone) immediately before PCI
* known intolerance to thiazolidinediones
* creatinine > 130 µmol/L
* significant liver disease: ALT or AST > 3 times upper limit of normal, history of cirrhosis, or hepatitis
* women who were pregnant, breastfeeding, or childbearing potential

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2002-08; Primary Completion 2006-11 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
The primary IVUS endpoint of the study was the change in three-dimensional neointimal plaque volume within the stented segment at follow-up, compared to baseline. | 6 months

SECONDARY OUTCOMES:
The secondary IVUS endpoint was the change in the two-dimensional NIA within the stent, using the cross-sectional slice showing the smallest LA on follow-up and comparing it to the corresponding baseline slice. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence M Title, MD FRCPC, Principal Investigator — QE II Health Sciences Centre
Locations (1):
- Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia, Canada